## Reducing Stigma towards Opioid Use Disorder on Interpersonal and Intrapersonal Levels

Statistical Analysis Plan

NCT04693416

12/7/2022

Preliminary data analyses will include studies of patterns of missing data, dropout rates, distributional properties of measures, and correlations among assessment measures. Continuous variables showing significant skewness or kurtosis will be analyzed with methods not sensitive to these features or will be transformed using standard approaches (such as Box-Cox transformations). Because all analyses will focus on feasibility and satisfaction and determining preliminary intervention effect sizes (with less concern focused on testing for statistical significance), outcome analyses will be conducted using a separate analysis for each outcome at the follow up observation.

Individual (intrapersonal) changes in stigma pre/post intervention will be conducted using paired sample t-test/Wilcoxon signed-rank test. Individual treatment uptake (agreement to set up an appointment and attendance at the appointment) will be included as secondary correlational analyses to evaluate relations with stigma scores. Comparisons with archival data will be conducted using a Chi Square analysis/Fisher's exact test. Family/Support (interpersonal) pre/post intervention outcomes will be conducted using paired sample t-test/Wilcoxon signed-rank test. Community assessment baseline and follow up data will be entered into a 2 (baseline vs. follow up) by 2 (intervention vs. comparison) analysis of variance (ANOVA) which will yield effect sizes for time, and interactions of time by intervention group. The primary dependent variable will be stigma score. We hypothesize that stigma scores will be lower in the intervention community.